CLINICAL TRIAL: NCT06484699
Title: Open Versus Laparoscopic Repair of Perforated Peptic Ulcer in Sohag
Brief Title: Open Versus Laparoscopic Repair of Perforated Peptic Ulcer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hussam Fathy Muhammad, Resident, Department of General Surgery, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-05-05MS
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-06

CONDITIONS: Perforated Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open repair of perforated peptic ulcer (Active Comparator): group (A) includes patients with perforated peptic ulcer that will be operated by open repair approach
  Interventions: Procedure: open repair of perforated peptic ulcer
- laparoscopic repair of perforated peptic ulcer (Active Comparator): group (B) includes patients with perforated peptic ulcer that will be operated by laparoscopic repair approach
  Interventions: Procedure: laparoscopic repair of perforated peptic ulcer

INTERVENTIONS:
Procedure: open repair of perforated peptic ulcer — group (A) includes patients with perforated peptic ulcer that will be operated by open repair approach
  Arms: open repair of perforated peptic ulcer
Procedure: laparoscopic repair of perforated peptic ulcer — group (B) includes patients with perforated peptic ulcer that will be operated by laparoscopic repair approach
  Arms: laparoscopic repair of perforated peptic ulcer

SUMMARY:
The aim of this clinical trial is to compare the outcomes of open versus laparoscopic repair for perforated peptic ulcer and provide evidence-based guidance to the selection of the most appropriate operative technique at Sohag University Hospital. The study will include patients presented with perforated peptic ulcers as a complication of peptic ulcer disease during the period of study.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a clinical diagnosis of perforated peptic ulcer that are fit to undergo surgery either via laparotomy or laparoscopy, males or females, any age, with gastric or duodenal ulcer, with American Society of Anesthesiologists (ASA) grade I, II, III.

Exclusion Criteria:

* Patients with associated bleeding ulcer (additional steps are needed to control bleeding).
* Patients with associated pathology other than perforated peptic ulcer.
* Patients with American Society of Anesthesiologists (ASA) grade IV, V, VI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Early postoperative follow up for repair of perforated peptic ulcer | 3 days after the operation
  resumption of oral intake

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Lanas A, Chan FKL. Peptic ulcer disease. Lancet. 2017 Aug 5;390(10094):613-624. doi: 10.1016/S0140-6736(16)32404-7. Epub 2017 Feb 25. PMID 28242110
- [Background] Tarasconi A, Coccolini F, Biffl WL, Tomasoni M, Ansaloni L, Picetti E, Molfino S, Shelat V, Cimbanassi S, Weber DG, Abu-Zidan FM, Campanile FC, Di Saverio S, Baiocchi GL, Casella C, Kelly MD, Kirkpatrick AW, Leppaniemi A, Moore EE, Peitzman A, Fraga GP, Ceresoli M, Maier RV, Wani I, Pattonieri V, Perrone G, Velmahos G, Sugrue M, Sartelli M, Kluger Y, Catena F. Perforated and bleeding peptic ulcer: WSES guidelines. World J Emerg Surg. 2020 Jan 7;15:3. doi: 10.1186/s13017-019-0283-9. eCollection 2020. PMID 31921329
- [Background] Lau JY, Sung J, Hill C, Henderson C, Howden CW, Metz DC. Systematic review of the epidemiology of complicated peptic ulcer disease: incidence, recurrence, risk factors and mortality. Digestion. 2011;84(2):102-13. doi: 10.1159/000323958. Epub 2011 Apr 14. PMID 21494041